CLINICAL TRIAL: NCT00445679
Title: A Multicenter, Randomized, Double-blind, Paroxetine-referenced, Parallel-group Study to Evaluate the Safety, Efficacy, and Tolerability of 3 Fixed Doses (50mg, 100mg, AND 200mg) of Desvenlafaxine Succinate Sustained-release Tablets in Adult Outpatients With Major Depressive Disorder
Brief Title: Paroxetine-referenced Study Evaluating Three Doses of DVS SR in Outpatients With MDD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3151A1-336
Record Dates: First submitted 2007-03-06; First posted 2007-03-09 (Estimated); Results first posted 2013-11-04 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-10

CONDITIONS: Depressive Disorder, Major
Keywords: major depressive disorder; MDD; depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Paroxetine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- A (Experimental): DVS SR 50mg/day
  Interventions: Drug: DVS SR
- B (Experimental): DVS SR 100mg/day
  Interventions: Drug: DVS SR
- C (Experimental): DVS SR 200mg/day
  Interventions: Drug: DVS SR
- D (Active Comparator): Paroxetine 20mg/day
  Interventions: Drug: Paroxetine

INTERVENTIONS:
Drug: DVS SR — Arm 1: 50mg DVS SR tablet, QD, 8 weeks treatment with 2 week taper Arm 2: 100mg DVS SR tablet, QD, 8 weeks treatment with 2 week taper Arm 3: 200mg DVS SR tablet, QD, 8 weeks treatment with 2 week taper
  Arms: A; B; C
Drug: Paroxetine — 20 mg Paroxetine capsule, QD, 8 weeks treatment with 2 week taper
  Arms: D

SUMMARY:
This study will assess the safety, tolerability and efficacy of desvenlafaxine succinate sustained release (DVS SR) in subjects with major depressive disorder.

DETAILED DESCRIPTION:
The primary objective of this study is to investigate the efficacy, safety and tolerability of desvenlafaxine succinate sustained release (DVS SR) in Chinese, Taiwanese, South Korean, and Indian subjects with major depressive disorder (MDD) receiving daily doses of 50 mg, 100 mg, or 200 mg. The secondary objective is to obtain additional information regarding the efficacy of DVS SR in subjects with MDD receiving daily doses of 50 mg, 100 mg, or 200 mg. Additional objectives include obtaining general and functional quality of life outcome data.

ELIGIBILITY:
Primary Inclusion Criteria:

1. Outpatient men and women at least 18 years of age.
2. Have a primary diagnosis of MDD based on the criteria in the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM IV), single or recurrent episode, without psychotic features.
3. Have a HAM D17 total score ≥20 at the screening and baseline (study day 1) visit.

Primary Exclusion Criteria:

1. Treatment with DVS SR at any time in the past.
2. Significant risk of suicide based on clinical judgment, including common suicidal thoughts and suicide having been considered as a possible solution even without specific plans or intent.
3. Any unstable hepatic, renal, pulmonary, cardiovascular (including uncontrolled hypertension), ophthalmologic, neurologic, or any other medical condition that might confound the study or put the subject at greater risk during study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 807 (Actual)
Dates: Start 2007-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For China: medinfo@wyeth.com
Locations (23):
- China (9):
  - Beijing
  - Guangdong Province
  - Hunan Province
  - Jiangsu Province
  - Shanghai
  - Shanxi Province
  - Sichuan Province
  - Yunnan Province
  - Zhejiang Province
- India (9):
  - Andhra Pradesh
  - Chandigarh
  - Gujarat
  - Karnataka
  - Maharashtra
  - Mumbai Maharashtra
  - New Delhi
  - Punjab
  - Uttar Pradesh
- South Korea (2):
  - Incheon
  - Seoul
- Taiwan (3):
  - Chang-hua
  - Kaohsiung City
  - Taipei

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in China, India, South Korea and Taiwan from July 2007 to December 2008.
Pre-assignment Details: After a 4 to 21 day screening period, eligible subjects were treated for up to 8 weeks.
Groups:
- DVS SR 50: Desvenlafaxine Succinate Sustained-Release (DVS SR) 50 mg/day
- DVS SR 100: Desvenlafaxine Succinate Sustained-Release (DVS SR) 100 mg/day
- DVS SR 200: Desvenlafaxine Succinate Sustained-Release (DVS SR) 200 mg/day
- Paroxetine 20: Paroxetine 20 mg/day
Period: Overall Study
Arm/Group | DVS SR 50 | DVS SR 100 | DVS SR 200 | Paroxetine 20
Started | 203 | 203 | 205 | 196
Completed | 155 | 157 | 139 | 149
Not Completed | 48 | 46 | 66 | 47
Not completed — Adverse Event | 22 | 12 | 30 | 19
Not completed — Failed to return | 1 | 3 | 2 | 2
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 10 | 6 | 6 | 5
Not completed — Compliance | 3 | 2 | 1 | 2
Not completed — Withdrawal of Informed Consent | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 2 | 3 | 3 | 1
Not completed — Withdrawal by Subject | 8 | 14 | 20 | 18
Not completed — Lack of Efficacy | 2 | 6 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DVS SR 50 | DVS SR 100 | DVS SR 200 | Paroxetine 20 | Total
Number analyzed (Participants) | 203 | 203 | 205 | 196 | 807
Age Continuous [Mean (Standard Deviation); unit: years] | 38.63 (12.96) | 39.26 (13.22) | 39.26 (14.69) | 38.27 (13.22) | 38.86 (13.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 129 | 118 | 117 | 489
  Male | 78 | 74 | 87 | 79 | 318

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders With a 50% or Greater Decrease From Baseline on the Hamilton Rating Scale for Depression, 17-item (HAM-D17)
Description: HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Items are scored on either a 3 point (0 to 2) or a 5 point scale (0 to 4), with 0=none/absent and 4=most severe, for a maximum total score of 50.
Time Frame: 8 weeks
Population: The intent-to-treat (ITT) population included all subjects randomly assigned to treatment who had a baseline HAM-D17 evaluation, took at least 1 dose of double-blind test article, and had at least 1 postbaseline HAM-D17 evaluation.
Measure: Number; unit: percentage of responders
Arm/Group | DVS SR 50 | DVS SR 100 | DVS SR 200 | Paroxetine 20
Number analyzed (Participants) | 200 | 200 | 197 | 192
percentage of responders | 63 | 67 | 63 | 66
Statistical Analysis 1: Comparison: DVS SR 50 vs Paroxetine 20; Test type: Non-Inferiority or Equivalence — Noninferiority to paroxetine was declared if the lower limit of the 95% two-sided confidence interval for the difference in responders is greater than or equal to -9 percentage points; Difference = -3.13, 95% CI 2-sided [-12.62 to 6.37]
Statistical Analysis 2: Comparison: DVS SR 100 vs Paroxetine 20; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.88, 95% CI 2-sided [-8.50 to 10.25]
Statistical Analysis 3: Comparison: DVS SR 200 vs Paroxetine 20; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -2.17, 95% CI 2-sided [-11.68 to 7.33]

2. Secondary Outcome: Clinical Global Impressions Scale-Improvement (CGI-I) Scores
Description: CGI-I is a global rating scale that measures disease improvement. Using a 7-point scale, the clinician rates how much the subject's illness has improved or worsened relative to the baseline status (1= very much improved; 7= very much worse).
Time Frame: 8 weeks
Population: The intent-to-treat (ITT) population included all subjects randomly assigned to treatment who had a baseline HAM-D17 evaluation, took at least 1 dose of double-blind test article, and had at least 1 postbaseline HAM-D17 evaluation. Number of participants analyzed reflects the final on-therapy population.
Measure: Number; unit: subjects
Arm/Group | DVS SR 50 | DVS SR 100 | DVS SR 200 | Paroxetine 20
Number analyzed (Participants) | 200 | 200 | 196 | 191
subjects
  Final - Score 1 (Very much improved) | 72 | 78 | 79 | 72
  Final - Score 2 (Much improved) | 64 | 64 | 53 | 59
  Final - Score 3 (Minimally improved) | 36 | 34 | 28 | 37
  Final - Score 4 (No change) | 16 | 17 | 26 | 17
  Final - Score 5 (Minimally worse) | 8 | 6 | 10 | 4
  Final - Score 6 (Much worse) | 4 | 1 | 0 | 2
  Final - Score 7 (Very Much worse) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: DVS SR 50 vs Paroxetine 20; Final on-therapy population; Test type: Superiority or Other; p = 0.714, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: DVS SR 100 vs Paroxetine 20; Final on-therapy population; Test type: Superiority or Other; p = 0.653, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: DVS SR 200 vs Paroxetine 20; Final on-therapy population; Test type: Superiority or Other; p = 0.881, Cochran-Mantel-Haenszel

3. Secondary Outcome: Clinical Global Impressions Scale-Severity of Illness (CGI-S) Scores
Description: CGI-S is a global rating scale that measures the severity of a subject's disease. Using a 7-point scale, the clinician rates the severity of the patient's mental illness at the time of the assessment, relative to the clinician's experience with subjects who have the same diagnosis (1= normal, not at all ill; 7= among the most extremely ill).
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | DVS SR 50 | DVS SR 100 | DVS SR 200 | Paroxetine 20
Number analyzed (Participants) | 200 | 200 | 197 | 192
subjects
  Final - Score 1 (Normal, not at all ill) | 40 | 50 | 53 | 42
  Final - Score 2 (Borderline mentally ill) | 49 | 53 | 47 | 49
  Final - Score 3 (Mildly ill) | 53 | 46 | 34 | 51
  Final - Score 4 (Moderately ill) | 29 | 30 | 38 | 27
  Final - Score 5 (Markedly ill) | 24 | 18 | 19 | 15
  Final - Score 6 (Severely ill) | 5 | 2 | 6 | 7
  Final - Score 7 (Among the most extremely ill) | 0 | 1 | 0 | 1
Statistical Analysis 1: Comparison: DVS SR 50 vs Paroxetine 20; Final on-therapy population; Test type: Superiority or Other; p = 0.450, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: DVS SR 100 vs Paroxetine 20; Final on-therapy population; Test type: Superiority or Other; p = 0.452, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: DVS SR 200 vs Paroxetine 20; Final on-therapy population; Test type: Superiority or Other; p = 0.850, Cochran-Mantel-Haenszel

4. Secondary Outcome: Montgomery and Asberg Depression Rating Scale (MADRS) Total Score Mean Change From Baseline
Description: Measures the overall severity of depressive symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Time Frame: Baseline and 8 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | DVS SR 50 | DVS SR 100 | DVS SR 200 | Paroxetine 20
Number analyzed (Participants) | 193 | 193 | 192 | 185
units on a scale | -16.84 [-18.37 to -15.31] | -17.84 [-19.37 to -16.31] | -16.81 [-18.43 to -15.20] | -16.54 [-18.08 to -15.00]

5. Secondary Outcome: Visual Analog Scale-pain Intensity (VAS-PI) Score Mean Change From Baseline
Description: The VAS-PI is a self-rated visual analog scale for the assessment of pain. Scores on the VAS-PI range from 0 (no pain) to 10 (worst possible pain). A decrease in VAS-PI overall scores indicates a subject's assessment of an improvement in pain.
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | DVS SR 50 | DVS SR 100 | DVS SR 200 | Paroxetine 20
Number analyzed (Participants) | 192 | 192 | 191 | 185
scores on a scale | -11.69 [-15.10 to -8.27] | -10.00 [-13.75 to -6.26] | -9.10 [-12.75 to -5.45] | -9.52 [-12.40 to -6.63]

6. Secondary Outcome: Hamilton Rating Scale for Depression, 6-item (HAM-D6) Score Mean Change From Baseline
Description: HAM-D6: standardized, clinician-administered rating scale is a subset of the HAM-D17 that assesses 6 items associated with major depression. The scale uses HAM-D17 items 1, 2, 7, 8, 10 and 13. Item 13 is scored 0 to 2 (0=none/absent to 2=most severe) and all others are scored 0 to 4 (0=none/absent to 4=most severe). Total score ranges from 0 to 22; higher score indicates more depression.
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | DVS SR 50 | DVS SR 100 | DVS SR 200 | Paroxetine 20
Number analyzed (Participants) | 200 | 200 | 197 | 192
scores on a scale | -6.50 [-7.08 to -5.92] | -6.51 [-7.06 to -5.95] | -6.42 [-7.03 to -5.82] | -6.58 [-7.15 to -6.01]

7. Secondary Outcome: Covi Anxiety Scale Score Mean Change From Baseline
Description: Covi anxiety scale measures the severity of anxiety symptoms on 3 items: verbal report, behavior and somatic complaints. Each dimension is assessed using a 5-point scale: 1 = not at all, 2 = somewhat, 3 = moderately, 4 = considerably, 5 = Very much. Total score ranges from 3 to 15; higher score indicates more anxiety.
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | DVS SR 50 | DVS SR 100 | DVS SR 200 | Paroxetine 20
Number analyzed (Participants) | 193 | 193 | 192 | 185
scores on a scale | -1.23 [-1.47 to -0.99] | -1.28 [-1.54 to -1.03] | -1.17 [-1.44 to -0.89] | -1.24 [-1.49 to -1.00]

ADVERSE EVENTS:
Arm/Group | DVS SR 50 | DVS SR 100 | DVS SR 200 | Paroxetine 20
Serious Adverse Events (participants affected / at risk) | 4/203 | 1/203 | 5/205 | 2/196
Other Adverse Events (participants affected / at risk) | 128/203 | 128/203 | 140/205 | 134/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DVS SR 50 (N=203) | DVS SR 100 (N=203) | DVS SR 200 (N=205) | Paroxetine 20 (N=196)
Cholelithiasis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pituitary tumor benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 2 | 0 | 2 | 1
Mania (Psychiatric disorders) | 1 | 0 | 1 | 0
Suicidal behavior (Psychiatric disorders) | 0 | 0 | 2 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 2
Drug abuse (Psychiatric disorders) | 0 | 0 | 0 | 1
Major Depressive Disorder worsening (Psychiatric disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DVS SR 50 (N=203) | DVS SR 100 (N=203) | DVS SR 200 (N=205) | Paroxetine 20 (N=196)
Palpitations (Cardiac disorders) | 9 | 7 | 12 | 10
Constipation (Gastrointestinal disorders) | 19 | 30 | 20 | 23
Dry mouth (Gastrointestinal disorders) | 17 | 16 | 19 | 12
Nausea (Gastrointestinal disorders) | 30 | 39 | 41 | 34
Asthenia (General disorders) | 8 | 5 | 11 | 6
Nasopharyngitis (Infections and infestations) | 5 | 8 | 11 | 13
Anorexia (Metabolism and nutrition disorders) | 13 | 14 | 12 | 14
Dizziness (Nervous system disorders) | 30 | 35 | 26 | 29
Headache (Nervous system disorders) | 17 | 20 | 16 | 14
Somnolence (Nervous system disorders) | 13 | 17 | 11 | 20
Insomnia (Psychiatric disorders) | 27 | 14 | 19 | 8
Dyspepsia (Gastrointestinal disorders) | 12 | 8 | 6 | 6
Sedation (Nervous system disorders) | 4 | 5 | 9 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.